CLINICAL TRIAL: NCT00816517
Title: Pilot Study on the Safety and Efficacy of Botulinum Toxin Injections in the Treatment of Psoriasis Vulgaris.
Brief Title: Use of Botulinum Toxin to Treat Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0808M45282
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis; Botulinum toxin
MeSH Terms: conditions — Psoriasis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- botulinum toxin (Experimental): injection of botulinum toxin type A
  Interventions: Biological: injection of botulinum toxin type A.

INTERVENTIONS:
Biological: injection of botulinum toxin type A. — 35 to 100 units injected around a skin lesion (plaque) one time.
  Other Names: Botox.

SUMMARY:
Psoriasis vulgaris is a chronic disease in which psoriatic plaques may appear on the knees, elbows, scalp and trunk. Evidence suggests the role of neurogenic inflammation in the pathogenesis of psoriasis. Botulinum toxin has been shown to have an effect on inhibiting neurogenic inflammation.

Recently, it was reported that patients who suffered from dystonia and had concomitant psoriasis, when treated with botulinum toxin for dystonia noted a dramatic improvement of their psoriatic lesions.

This pilot study will determine the safety and efficacy of botulinum toxin in the management of psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects. Psoriasis vulgaris diagnosis made by a board certified dermatologist involving at least one area that has been intolerant or recalcitrant to at least two forms of recognized topical or systemic treatments in the past. In addition, the subject should have at least a score of 2 for keratoderma and erythema. Signed informed consent. Willing to adhere to protocol.

Exclusion Criteria:

* Immunosuppressed patients, pregnant, secondary skin infections, phototherapy within 4 weeks of the botulinum toxin injection, exposure to any topical or systemic retinoid treatment with the last 12 months, volunteers taking chloroquine and hydroxychloroquine, volunteers on warfarin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
psoriasis scoring scale | baseline and 3months

SECONDARY OUTCOMES:
3mm skin biopsy. | baseline and at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- Univerisity of Minnesota, Minneapolis, Minnesota, United States